CLINICAL TRIAL: NCT04193319
Title: Study on the Pharmacokinetics of Fluconazole on Single-center, One-arm, Open and Fixed Sequences of Fluzoparib in Healthy Male Subjects
Brief Title: Effect of Fluconazole on PK of Fluzoparib in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FZPL-I-108
Record Dates: First submitted 2019-11-21; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — fluzoparib; Fluconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other)
  Interventions: Drug: Fluzoparib; Drug: Fluconazole

INTERVENTIONS:
Drug: Fluzoparib — PARP inhibitor
Drug: Fluconazole — inhibitor

SUMMARY:
The purpose of this study is to evaluate the Effect of fluconazole on the Pharmacokinetics of Fluzoparib in Healthy male Adults

DETAILED DESCRIPTION:
Subjects received oral Fluzoparib 20 mg after D1 single meal, D2-D4 for washing period, D5 started oral fluconazole 400 mg/day/day after meal, continuous administration for 6 days to D10, D8 meal After oral administration of fluconazole 400 mg, a single oral dose of Fluzoparib 20 mg was given immediately.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 35- 50 years old (including both ends), male;
2. The body weight is not less than 50 kg, and the body mass index [BMI = weight kg / (height m) 2] is in the range of 18 to 28 (including the critical value);
3. Subjects are willing to have no birth plans in the next 6 months and voluntarily take effective contraceptive measures;
4. Good health, no history of heart, liver, kidney, digestive tract, nervous system and metabolic abnormalities;
5. There are no abnormalities or abnormalities in vital signs and physical examination.
6. Understand the research procedures and methods, voluntarily participate in the trial, and sign the informed consent in writing. Fully understand the test content, process and possible adverse reactions;
7. Creatinine is less than or equal to the upper limit of normal;

Exclusion Criteria:

1. Participate in blood donation within 3 months before screening and donate blood volume ≥400mL or blood loss ≥400mL, participate in blood donation within one month and donate blood volume ≥200mL or blood loss ≥200mL, or receive blood transfusion;
2. Allergies, including a history of severe drug allergies or drug allergies; a history of allergies to fluzolidine capsules or their excipients.
3. Those who have a history of drug and/or alcohol abuse, who are positive for alcohol and drug screening, or who have used drug abuse in the past five years or who have used drugs three months before the test;
4. People who smoke alcohol (drinking 14 units of alcohol per week: 1 unit = beer 285 mL, or spirits 25 mL, or wine 100 mL; daily smoking ≥ 5) and can not be smoke-free and alcohol-free during the test period ;
5. Those with previous history of cardiovascular disease such as cardiac insufficiency, myocarditis, coronary heart disease, pathological arrhythmia, and stroke;
6. Pulmonary diseases, including invasive lung disease, pneumonia, difficulty breathing, etc.;
7. History of chronic kidney disease, renal insufficiency, and renal anemia;
8. Have a history of dysphagia or any history of gastrointestinal disease that affects drug absorption;
9. Any uncontrolled peptic ulcer, inflammatory bowel disease, pancreatitis, etc.;
10. Anyone who has undergone any surgery within the first 6 months of screening; has undergone any surgery that affects gastrointestinal absorption (including gastrectomy, bowel resection, stomach reduction, etc.)
11. A clear history of other major organ diseases such as the nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and musculoskeletal system within the first month prior to screening (eg uncontrolled diabetes, hypertension) Etc.), making the researcher feel unsuitable for participation in the study;
12. Hepatotoxic drugs (such as acetaminophen, statin lipid-lowering drugs, azithromycin, dapsone, clarithromycin, fluconazole, ketoconazole, etc. within 6 months prior to screening (for more than 2 consecutive weeks) Li Fuping);
13. Those who have taken any clinical trial drug within 3 months;
14. Take any medication that alters liver enzyme activity 28 days prior to taking the study drug (see Appendix 1);
15. Take any prescription or over-the-counter medication 14 days before taking the study drug;
16. Ingested any vitamin products or herbs 14 days prior to taking the study drug;
17. Clinical laboratory tests are abnormal and clinically significant, or other clinical findings indicate the following diseases (including but not limited to gastrointestinal, renal, hepatic, neurological, blood, endocrine, tumor, lung, immune, mental or cardiovascular) disease);
18. Concomitant infection with other viruses (anti-HCV, anti-HIV positive, HBsAg positive) or syphilis infection;
19. Ingested grapefruit or grapefruit-containing products, caffeine, jaundice or alcoholic foods or beverages (including chocolate, tea, coffee, cola, etc.) 48 hours prior to taking the study drug; strenuous exercise, or other Factors affecting drug absorption, distribution, metabolism, excretion, etc.;
20. According to the chest X-ray and abdominal B-ultrasound examination items at the time of screening, abnormalities and clinical significance were confirmed.
21. The investigator believes that there are other subjects who are not eligible to participate in this trial.

Ages: 35 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration(Cmax) of Fluzoparib | through study completion，up to 24 weeks
  Cmax
Area under the Plasma Concentration-time curve From 0-t of Fluzoparib | through study completion，up to 24 weeks
  AUC0-t
Area under the Plasma Concentration-time curve From 0 to infinity of Fluzoparib | through study completion，up to 24 weeks
  AUC0-∞

SECONDARY OUTCOMES:
Safety in terms of Adverse Events Assessments | through study completion，up to 24 weeks
  NCI-CTC AE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Early Cancer Research Center of Hunan Cancer Hospital, Hunan, Hunan, China